CLINICAL TRIAL: NCT07140406
Title: Three-dimensional Motion Capture System Combined With sEMG Was Used to Evaluate the Effect of Different Firebone Acupuncture Strategies on Upper Limb Function in Stroke Patients
Brief Title: Observation of the Therapeutic Effect of Fire Needle on Upper Limb Function in Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, ZhangZhaohui, Acupuncture and moxibustion therapist, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202309-045-2
Record Dates: First submitted 2025-07-28; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Infarction
Keywords: dysfunction; stroke; fire needle; Surface electromyography; 3D motion capture system
MeSH Terms: conditions — Cerebral Infarction; Stroke | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Flexed muscle Milli-fire needle (Experimental): Patients in the flexor treatment group received conventional rehabilitation training, conventional acupuncture, and moxibustion with fine fire needles on the flexor muscle groups (biceps brachii and forearm flexor muscle groups).The Milli-fire needle treatment was administered every other day for a total of 4 weeks.
  Interventions: Other: conventional rehabilitation training; Other: conventional acupuncture; Other: Acupuncture with the milli-needle fire-puncture on flexor muscle groups
- Extensor muscle Milli-fire needle (Experimental): The patients in the extensor muscle treatment group received conventional rehabilitation training , conventional acupuncture and moxibustion with Milli-fire needle on the extensor muscle groups (triceps brachii, forearm extensor muscles).The Milli-fire needle treatment was administered every other day for a total of 4 weeks.
  Interventions: Other: conventional rehabilitation training; Other: conventional acupuncture; Other: Acupuncture with the milli-needle fire-puncture on extensor muscle groups
- Control group (Active Comparator): Patients in the control group received conventional rehabilitation training, conventional acupuncture, and conventional moxibustion with Milli-fire needle.The acupuncture points for fire needle puncture are commonly used ones on the upper limbs.The Milli-fire needle treatment was administered every other day for a total of 4 weeks.
  Interventions: Other: conventional rehabilitation training; Other: conventional acupuncture; Other: Conventional needle puncture with a fire needle

INTERVENTIONS:
Other: conventional rehabilitation training — The rehabilitation training is designed based on the specific functional conditions of the patient's limbs. The specific training methods include proper limb positioning, exercise therapy such as passive movement, anti-spasticity training, scapular girdle muscle training, joint extension training, forearm pronation and supination training, occupational therapy, joint movement training, roller treatment, and fine motor skill training, etc. The treatment is conducted once a day and five times a week. The treatment lasts for 4 consecutive weeks.
Other: conventional acupuncture — Conventional acupuncture treatment involves needling at acupoints on the upper limbs of patients to improve their upper limb function. The treatment is administered once a day, five times a week, for a continuous period of four weeks.
Other: Acupuncture with the milli-needle fire-puncture on flexor muscle groups — The acupuncture points of the milli-needle fire-puncture device are located in the flexor muscle groups of the upper limbs, including the biceps brachii and the flexor muscle group of the forearm.
  Arms: Flexed muscle Milli-fire needle
Other: Acupuncture with the milli-needle fire-puncture on extensor muscle groups — The acupuncture points for the milli-needle fire-puncture device are located in the extensor muscle groups of the upper limbs, including the triceps brachii and the extensor muscles of the forearm.
  Arms: Extensor muscle Milli-fire needle
Other: Conventional needle puncture with a fire needle — The acupuncture points for milli-needle fire-puncture are commonly used ones on the upper limbs.
  Arms: Control group

SUMMARY:
Objective: To explore the clinical efficacy of different needling strategies with moxibustion needles on upper limb function in post-stroke patients. Method: 105 patients with upper limb dysfunction after stroke were randomly divided into an extensor treatment group, a flexor treatment group, and a control group, with 35 patients in each group. Patients in the extensor treatment group were treated with extensor group moxibustion, patients in the flexor treatment group were treated with flexor group moxibustion, and patients in the control group were treated with conventional moxibustion. Observe the upper limb movement trajectory, surface electromyographic signals (sEMG) of extensor and flexor muscle groups, MAS scale scores, and FMA-UE scores of two groups of patients under specific tasks detected by a three-dimensional motion capture system before and after treatment, and determine the clinical efficacy. Result: Moxibustion therapy with moxibustion is helpful in improving upper limb dysfunction in stroke patients, safe and reliable, and worthy of application. The efficacy of needling the flexor muscle group with moxibustion is better than that of needling the extensor muscle group and conventional acupuncture, providing certain evidence and guidance for the selection of moxibustion sites in clinical practice.

DETAILED DESCRIPTION:
105 patients with upper limb dysfunction after stroke were selected according to the inclusion criteria and randomly divided into an extensor treatment group, a flexor treatment group, and a control group of 35 cases each. The patients in the extensor treatment group were treated with routine rehabilitation training+routine acupuncture and moxibustion+millifire needle acupuncture for the extensor muscle group (triceps brachii, forearm extensor muscle group), the patients in the flexor treatment group were treated with routine rehabilitation training+routine acupuncture and moxibustion+millifire needle acupuncture for the flexor muscle group (biceps brachii, forearm flexor muscle group), and the patients in the control group were treated with routine rehabilitation training+routine acupuncture and moxibustion+routine millifire needle acupuncture. The treatment was administered once every other day with a moxibustion needle for a total of 4 weeks. Observe the upper limb movement trajectory, surface electromyographic signals (sEMG) of extensor and flexor muscle groups, changes in MAS scale scores, and FMA-UE scores of two groups of patients under specific tasks detected by a three-dimensional motion capture system before, after one treatment, and after 4 weeks of treatment. Calculate joint angles and motion distances through spatial coordinates, and apply RMS MF、CC、 Coherence analysis quantifies muscle strength, muscle tension, fatigue, and coordination.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria.
2. The patient had a first stroke and the course of disease was 15 days to 12 months.
3. With unilateral disease， the muscular tone assessed by the modified Ashworth scale of upper limb was Ⅰ/Ⅰ+/Ⅱ/Ⅲ level ，Brunnstrom stage in upper limb was Ⅲ/Ⅳ/Ⅴ， Upper limb muscle strength is greater than or equal to grade 2.
4. Age 18-70 years old.
5. Have not taken Chinese or Western medicine sedatives muscle relaxants or any drugs that have an impact on muscle tone recently.
6. Clear consciousness stable vital signs no other acute diseases and serious complications.
7. Patients or family members agree to accept this clinical study and have signed informed consent.

Exclusion Criteria:

1. Bilateral disease.
2. History of serious injury or disease of other upper limb nerves muscles or bones.
3. Patients with severe cervical spondylosis and hypertension.
4. Patients with audiovisual abnormalities severe cognitive impairment and mental diseases who cannot cooperate with the examination.
5. Patients with tumor and severe malnutrition.
6. There are contraindications for needle treatment such as extreme hunger tension infectious diseases skin collapse etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-12-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Root mean square(RMS) of surface electromyography(sEMG） | 4 weeks
  Using sEMG the EMG of the upper limb muscles is collected including RMS

SECONDARY OUTCOMES:
RMS of sEMG | first day
  Using sEMG, the EMG signals of the upper limb muscles are collected, including RMS .
Mean Frequency (MF)of SEMG | first day
  Using sEMG, the EMG signals of the upper limb muscles are collected, including MF.
Joint angle | first day
  Three-dimensional motion capture system was used to detect joint angle .
Motion distance | first day
  Three-dimensional motion capture system was used to detect motion distance.
Joint angle | 4 weeks
  Three-dimensional motion capture system was used to detect joint angle .
Motion distance | 4 weeks
  Three-dimensional motion capture system was used to detect motion distance.
Fugl-Meyer Assessment Upper Extremity Scale(FMA-UE) | 4 weeks
  FMA-UE is a commonly used scale for assessing upper limb motor function in stroke patients, mainly evaluating reflex activity, motor control, and muscle strength of the hemiplegic upper limb. FMA-UE includes 33 items related to proximal and distal limb movements of the upper limbs, with each item scored on a scale of 0, 1, and 2. 0 points indicates complete inability to complete, 2 points indicates ability to complete the specified action, and 1 point falls between the two; The total score ranges from 0 to 66 points. The higher the score, the better the upper limb function.
Modified Ashworth Scale(MAS) | 4 weeks
  MAS is a standardized tool for assessing the degree of muscle spasms and has been established as the clinical gold standard in the assessment of limb spasms after stroke. This scale is divided into levels 0-4, with higher levels indicating greater muscle tone.
Mean Frequency (MF)of SEMG | 4 weeks
  Using sEMG, the EMG signals of the upper limb muscles are collected, including MF.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
The original data will be released on 2026.12.30,and the method will be dislosed through the publishde papers.
Supporting Information: Study Protocol, SAP, ICF, CSR